CLINICAL TRIAL: NCT02338830
Title: Vaginal Progesterone for Prevention of Preterm Labor in Asymptomatic Twin Pregnancies With Sonographic Short Cervix
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mohamed Sayed Abdelhafez (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Abdelhafez, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WR1
Record Dates: First submitted 2014-12-24; First posted 2015-01-14 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Premature Labour
Keywords: Twins; Preterm labor; Progesterone; Short cervix
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progesterone group (Active Comparator): Women received vaginal progesterone suppositories
  Interventions: Drug: Progesterone
- No treatment group (No Intervention): Women received no treatment

INTERVENTIONS:
Drug: Progesterone — Women received vaginal progesterone suppositories (Cyclogest®, Actavis, Barnstaple, EX32 8NS, United Kingdom) in a dose of 400 mg daily beginning at 20-24 weeks gestational age
  Other Names: Cyclogest
  Arms: Progesterone group

SUMMARY:
To evaluate the value of vaginal progesterone therapy for reduction of preterm labor in asymptomatic twin pregnancies who have sonographic short cervix

DETAILED DESCRIPTION:
Women with twin pregnancy with transvaginal sonographic cervical length of 20-25 mm at 20-24 weeks gestational age without symptoms, signs or other risk factors of preterm labor will be included in the study. All women will be randomly divided into two groups; one group (study group) received vaginal progesterone suppositories in a dose of 400 mg daily beginning at 20-24 weeks gestational age (study group) and the other group received no treatment (control group)

ELIGIBILITY:
Inclusion Criteria:

* Women pregnant in dichorionic twins.
* Transvaginal sonographic cervical length is 20-25 mm at 20-24 weeks gestational age.
* No symptoms, signs or other risk factors for preterm labor.

Exclusion Criteria:

* Age < 20 years or > 35 years.
* Known allergy or contraindication (relative or absolute) to progesterone therapy.
* Pregnancy by in vitro fertilization (IVF) / intracytoplasmic sperm injection (ICSI).
* Monochorionic twins.
* Known major fetal structural or chromosomal abnormality.
* Intrauterine death of one fetus or death of both fetuses.
* Fetal reduction in current pregnancy.
* Cervical cerclage in current pregnancy.
* Medical conditions that may lead to preterm delivery.
* Rupture of membranes.
* Vaginal bleeding.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 182 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Preterm labor before 34 weeks | Up to 34 weeks gestational age

SECONDARY OUTCOMES:
Neonatal respiratory distress syndrome (RDS) | At birth
Early neonatal death (END). | One month after birth

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-refaie, Dr, Principal Investigator — Mansoura University; Mohamed S Abdelhafez, Dr, Study Director — Mansoura University; Ahmed M Badawy, Prof, Study Chair — Mansoura University
Locations (2):
- Egypt (2):
  - Obstetrics and Gynecology Department in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Private practice settings, Al Mansurah, Dakahlia Governorate